CLINICAL TRIAL: NCT01265472
Title: Comparison of the Expression Level of Translocator Protein (TSPO) and Binding Activity in Normal Cutaneous Tissue Versus Non Melanotic Cutaneous Malignancy.
Brief Title: Comparison of Translocator Protein Expression and Binding Activity in Normal Tissue Versus Non Melanotic Malignancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Rafael Nagler, Rambam Health Care Campus
Other Study IDs: RMB455-CTIL
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: Translocator Protein; Basal Cell Carcinoma; Squamous Cell Carcinoma; Malignancy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Basal Cell; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens of normal skin, squamous cell carcinoma or basal cell carcinoma
Oversight: Data Monitoring Committee: No

SUMMARY:
Translocator protein (TSPO) is a intracellular protein that is found primarily in the outer membrane of the mitochondria that is encoded by the TSPO gene. It has been found that TSPO expression in the skin correlates with cell proliferation and differentiation. Many studies have shown that TSPO overexpression in solid malignancies such as in ovarian cancer, colon cancer, and others, was also found to correlate with more aggressive cancer behavior. Working Hypothesis and Aims: Previous studies described an aberrant expression of TSPO levels in solid malignancies as compared to normal tissues. It is assumed that this aberration can be found in cuntaneous malignancies as well. The occurrence of this aberration may lead to the understanding of the mechanism of TSPO involment in the cutaneous malignancy, and in malignancies in general. Methods: The study will be carried out on surgically resected skin lesions suspected to SCC or BCC, which will be removed as part of the surgical routine treatment. The excision will be made in elliptic shape including the lesion and a part of normal skin surrounding it. A sample will be taken from the central part of the lesion and from the external extremity of the normal tissue. Western Blot will be conducted to detect the expression of TSPO. Binding activity with the TSPO specific ligandwill also be determined. Expected Results: We expect to observe either (a) a higher level of TSPO expression and a lower binding activity in malignant tissue compared with healthy control tissue or (b) a higher level of TSPO expression and a lower binding activity in malignant tissue compared with healthy control tissue. Importance: Until today, only a very small number of studies have examined TSPO in cutaneous malignancies, and these only examined TSPO expression. Our study will also measure the binding activity of TSPO in cutaneous malignant tissues compared to normal tissues

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Basal Cell Carcinoma or Squamous Cell Carcinoma

Exclusion Criteria:

* Non-compliance with inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Not an observational study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)